CLINICAL TRIAL: NCT04075682
Title: Evaluation of Cigarette Package Inserts for Enhanced Communication With Smokers
Brief Title: Cigarette Pack Inserts for Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: Cornell University (Other); University of Waterloo (Other); University of Tasmania (Other)
Responsible Party: Principal Investigator, James Francis Thrasher, PhD, Professor, University of South Carolina
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00083728
Record Dates: First submitted 2019-08-20; First posted 2019-09-03 (Actual); Results first posted 2024-05-13 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2023-11

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Intervention Model Description: In a 2 X 2 between subject design, smokers will be randomized into one of four cigarette package labeling conditions: 1. no inserts or pictorial HWLs; 2. inserts only; 3. pictorial HWLs only; 4. inserts & pictorial HWLs
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard cigarette packs (control) (No Intervention): Participants will be provided with a 2 week supply of their preferred brand of cigarettes, with the only alteration being the small health warning message on the side of the pack, whose textual content will be the same as that used for the pictorial warning label conditions.
- Cigarette packs with inserts only (Experimental): Participants will be provided with a 2 week supply of their preferred brand of cigarettes, with packs altered to include inserts with four different rotating messages to promote response efficacy beliefs (2 inserts on the benefits of cessation) or self-efficacy to quit (2 inserts with cessation tips).
  Interventions: Other: Inserts with efficacy messages
- Cigarette packs with pictorial warnings only (Experimental): Participants will be provided with a 2 week supply of their preferred brand of cigarettes, with packs altered to include four different rotating pictorial warnings showing the consequences of smoking and that cover 50% of the front and back of the pack.
  Interventions: Other: Pictorial warnings on packs
- Cigarette packs with inserts and pictorial warnings (Experimental): Participants will be provided with a 2 week supply of their preferred brand of cigarettes, with packs altered to include inserts with four rotating efficacy messages (see description above) and four rotating pictorial warnings (see above).
  Interventions: Other: Inserts with efficacy messages; Other: Pictorial warnings on packs

INTERVENTIONS:
Other: Inserts with efficacy messages — Four rotating inserts (i.e., small, printed messages) with messages about cessation benefits (i.e., response efficacy) and tips to quit (i.e., self-efficacy messages) will be placed inside cigarette packs.
  Arms: Cigarette packs with inserts and pictorial warnings; Cigarette packs with inserts only
Other: Pictorial warnings on packs — Four rotating pictorial warnings illustrating the harms of smoking will be printed on labels that will placed on and cover approximately 50% of the cigarette packs.
  Arms: Cigarette packs with inserts and pictorial warnings; Cigarette packs with pictorial warnings only

SUMMARY:
This study will test whether cigarette package inserts (i.e., small printed leaflets inside cigarette packs) with messages about the benefits of cessation and tips for quitting can help smokers quit. To do this, the investigators will conduct a 2 X 2 between-subject experiment in which 380 smokers will be randomized into one of four labeling groups: 1. no inserts or pictorial health warning labels (HWLs); 2. inserts only; 3. pictorial HWLs only; 4. inserts & pictorial HWLs. Smokers will be given a 14-day supply of their preferred cigarette brand with packs labeled according to their experimental group. Participants will answer a brief survey at the end of each day and four other times each day, using ecological momentary assessment approaches. The investigators will study whether smokers in each group experience different psychological responses and behaviors associated with smoking cessation.

ELIGIBILITY:
Inclusion Criteria:

* 18 or older
* Have smoked at least 100 cigarettes in their lifetime
* Smoked at least 10 cigarettes a day in the prior month.

Exclusion Criteria:

* Use of other nicotine products besides cigarettes in the prior month.
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 387 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2021-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James F Thrasher, PhD, Principal Investigator — University of South Carolina
Locations (2):
- United States (2):
  - Cornell University, Ithaca, New York
  - University of South Carolina, Columbia, South Carolina

IPD SHARING:
Plan to Share IPD: No
We are likely to make participant data to researchers who make specific requests and have specific data analysis plans that we approve.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Cigarette Packs (Control) | Cigarette Packs With Inserts Only | Cigarette Packs With Pictorial Warnings Only | Cigarette Packs With Inserts and Pictorial Warnings
Started | 108 | 94 | 94 | 91
Completed | 101 | 87 | 90 | 89
Not Completed | 7 | 7 | 4 | 2
Not completed — Lost to Follow-up | 5 | 5 | 2 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 1 | 0
Not completed — Not literate enough to self-administer study surveys | 1 | 0 | 0 | 0
Not completed — Lost study phone the first day of study participation | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The analysis population is those participants who were included in the analytic sample.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Cigarette Packs (Control) | Cigarette Packs With Inserts Only | Cigarette Packs With Pictorial Warnings Only | Cigarette Packs With Inserts and Pictorial Warnings | Total
Number analyzed (Participants) | 101 | 87 | 90 | 89 | 367
Age, Customized [Count of Participants; unit: Participants]
  18-35 years old | 27 | 27 | 26 | 21 | 101
  36-55 years old | 54 | 42 | 46 | 49 | 191
  56 years old and older | 20 | 18 | 18 | 19 | 75
Sex: Female, Male [Count of Participants; unit: Participants]
  Sex: Female | 60 | 52 | 52 | 61 | 225
  Sex: Male | 41 | 35 | 38 | 28 | 142
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 0 | 1 | 4
  Asian | 1 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  Black or African American | 17 | 8 | 8 | 14 | 47
  White | 75 | 74 | 73 | 71 | 293
  More than one race | 2 | 2 | 3 | 1 | 8
  Unknown or Not Reported | 4 | 2 | 4 | 2 | 12
Region of Enrollment [Number; unit: participants]
  United States | 101 | 87 | 90 | 89 | 367
Educational Attainment [Number; unit: participants] — This measure is the dichotomized version of our original question and is what we used when assessing moderation of insert effects (H6a, H6b).
  participants
    High School Education or less | 48 | 36 | 30 | 39 | 153
    Greater than High School Education | 53 | 49 | 57 | 50 | 209
    Missing | 0 | 2 | 3 | 0 | 5
Health Literacy [Number; unit: participants] — Health Literacy was assessed with the 6-item Newest Vital Sign, which categorizes people as having adequate, possibly limited or limited health literacy. For our assessment of moderation of insert effects by health literacy (i.e., H6a, H6b), we created a dichotomous measure by combining the categories of possibly limited or limited.
  participants
    Adequate | 66 | 61 | 66 | 63 | 256
    Limited OR Possibly Limited | 35 | 26 | 24 | 26 | 111
Self-efficacy to quit smoking [Mean (Standard Deviation); unit: units on a scale] — Population: This 3-item scale with Likert response options was averaged across the three items and has a range of 1-5, where higher values represent a better outcome (i.e., greater confidence to quit smoking).
  units on a scale
    number analyzed (Participants) | 100 | 83 | 88 | 88 | 359
    (all) | 2.32 (1.06) | 2.30 (0.92) | 2.39 (1.05) | 2.21 (0.81) | 2.31 (0.97)
Delayed Discounting [Mean (Standard Deviation); unit: units on a scale] — This measure assessed valuation of present rewards over future rewards, in which participants answer 5 questions with branching logic. Final values range from .0001 to 24 with a median of .0095, which we used to classify participants as having high vs. low delayed discounting. Low delayed discounting is indicative of a "better" outcome because people classified in this group are more likely to value future rewards (e.g., living longer) over present rewards (e.g., nicotine dosing), whereas the opposite is true for those with high delayed discounting.
  units on a scale | 0.56 (3.37) | 0.40 (2.70) | 0.36 (2.56) | 0.60 (3.57) | 0.48 (3.08)

OUTCOME MEASURES:

1. Primary Outcome: Self-efficacy to Quit Smoking
Description: A single question measured on a continuous scale (1="Not at all", worse outcome; 7="Extremely", better outcome) to assess strength of confidence to quit smoking, with average scores (range 1-7) estimated.
Time Frame: Evaluated approximately 4-5 times a day over the 14 day study period, with analyses limited to days 2-14. Day 1 was dropped due to varying coverage of the day depending on study orientation time.
Population: Analyses include repeated observations from daily cigarette surveys. Analytic samples for H6 differ due to some missing data for each moderating variable: education (control=101; insert only=84; pictorial warnings only=87; insert + pictorial warnings=88); health literacy (control=101; insert only=86; pictorial warnings only=90; insert + pictorial warnings=88); and delayed discounting (control=101; insert only=84; pictorial warnings only=88; insert + pictorial warnings=88).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Cigarette Packs (Control) | Cigarette Packs With Inserts Only | Cigarette Packs With Pictorial Warnings Only | Cigarette Packs With Inserts and Pictorial Warnings
Number analyzed (Participants) | 101 | 86 | 90 | 89
score on a scale | 2.61 (1.44) | 2.76 (1.55) | 2.62 (1.52) | 2.56 (1.40)
Statistical Analysis 1: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; These results are for the pre-specified H1 assessment (see Statistical Analysis Plan, Model 1), comparing groups that received inserts (insert only AND insert + pictorial warnings) with the groups that did not (pictorial warning only AND control). We expected that the outcome would be higher in the insert groups than in the no insert groups; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus their not being equal; p = 0.60, Mixed Models Analysis — The reported p-value is not adjusted. The a priori threshold for statistical significance uses a Bonferroni-adjusted critical value of p<0.05/6=0.0083; We estimated mixed-effects ordinal regression models that accounted for repeated measures at both the day- and individual-levels; Mean Difference (Net) = 0.26, 95% CI 2-sided [-0.73 to 1.25], Standard Error of Mean 0.51 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 2: Comparison: Cigarette Packs With Inserts Only vs Cigarette Packs With Inserts and Pictorial Warnings; These results are for the pre-specified H3 assessment (see Statistical Analysis Plan, Model 1), comparing the group that received inserts and pictorial warnings with the group that received inserts only. We expected that this outcome would be higher in the insert and pictorial warning group than in the insert only group; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus their not being equal; p = 0.29, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.78, 95% CI 2-sided [-2.22 to 0.66], Standard Error of Mean 0.73 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 3: Comparison: Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; These results are for the pre-specified H4 assessment (see Statistical Analysis Plan, Model 1), comparing the group that received inserts and pictorial warnings with the group that received pictorial warnings only. We expected that this outcome would be higher in the insert and pictorial warning group than in the pictorial warning only group; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.73, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.25, 95% CI 2-sided [-1.67 to 1.16], Standard Error of Mean 0.72 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 4: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; These results are for the intended (but not correctly pre-specified) H6a assessment, which evaluates moderation of the pre-specified H1 assessment. We expected that the effect of inserts (averaged over pictorial warnings) compared to no inserts (averaged over pictorial warnings) on the outcome would be stronger for those with higher than lower education (see Statistical Analysis Plan, Model 5); Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.77, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.30, 95% CI 2-sided [-2.34 to 1.74], Standard Error of Mean 1.04 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 5: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; These results are for the intended (but not correctly pre-specified) H6a assessment, which evaluates moderation of the pre-specified H1 assessment. We expected that the effect of inserts (averaged over pictorial warnings) compared to no inserts (averaged over pictorial warnings) on the outcome would be stronger for those with higher than lower literacy (see Statistical Analysis Plan, Model 5); Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.51, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.73, 95% CI 2-sided [-1.43 to 2.88], Standard Error of Mean 1.10 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 6: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; These results are for the intended (but not correctly pre-specified) H6a assessment, which evaluates moderation of the pre-specified H1 assessment. We expected that the effect of inserts (averaged over pictorial warnings) compared to no inserts (averaged over pictorial warnings) on the outcome would be stronger for those with lower than higher delayed discounting (see Statistical Analysis Plan, Model 5); Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.05, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 2.02, 95% CI 2-sided [0.02 to 4.01], Standard Error of Mean 1.02 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 7: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Inserts and Pictorial Warnings; These results are for the intended (but not correctly pre-specified) H6b assessment, which evaluated whether the moderation of insert effects would vary by whether the inserts included pictorial warnings or not. We expected that moderation by baseline education would be stronger for insert only (vs control) than for inserts AND pictorial warnings (vs control) (see Statistical Analysis Plan, Model 5); Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.54, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.91, 95% CI 2-sided [-3.84 to 2.02], Standard Error of Mean 1.49 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 8: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Inserts and Pictorial Warnings; These results are for the intended (but not correctly pre-specified) H6b assessment, which evaluated whether the moderation of insert effects would vary by whether the inserts included pictorial warnings or not. We expected that moderation by baseline literacy would be larger for insert only (vs control) than for inserts AND pictorial warnings (vs control) (see Statistical Analysis Plan, Model 5); Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.21, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 2.02, 95% CI 2-sided [-1.13 to 5.17], Standard Error of Mean 1.61 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 9: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Inserts and Pictorial Warnings; These results are for the intended (but not correctly pre-specified) H6b assessment, which evaluated whether the moderation of insert effects would vary by whether the inserts included pictorial warnings or not. We expected that moderation by baseline delay discounting would be larger for insert only (vs control) than for inserts AND pictorial warnings (vs control) (see Statistical Analysis Plan, Model 5); Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.47, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -1.07, 95% CI 2-sided [-3.97 to 1.83], Standard Error of Mean 1.48 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter

2. Primary Outcome: Self-efficacy to Cut Down on Smoking
Description: A single question measured on a continuous scale (1="Not at all", worse outcome; 7="Extremely", better outcome) to assess strength of confidence to cut down on the number of cigarettes smoked, with average scores (range=1-7) estimated.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Cigarette Packs (Control) | Cigarette Packs With Inserts Only | Cigarette Packs With Pictorial Warnings Only | Cigarette Packs With Inserts and Pictorial Warnings
Number analyzed (Participants) | 101 | 86 | 90 | 89
score on a scale | 3.15 (1.42) | 3.52 (1.59) | 3.29 (1.51) | 3.18 (1.56)
Statistical Analysis 1: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 1]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.57, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.28, 95% CI 2-sided [-0.68 to 1.24], Standard Error of Mean 0.49 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 2: Comparison: Cigarette Packs With Inserts Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 2]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.08, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -1.25, 95% CI 2-sided [-2.63 to 0.14], Standard Error of Mean 0.71 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 3: Comparison: Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; These results are for the pre-specified H4 assessment, comparing the group that received inserts and pictorial warnings with the group that received pictorial warnings only. We expected that this outcome would be higher in the insert and pictorial warning group than in the pictorial warning only group; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.39, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.60, 95% CI 2-sided [-1.97 to 0.77], Standard Error of Mean 0.70 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 4: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 4]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.61, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.51, 95% CI 2-sided [-1.45 to 2.47], Standard Error of Mean 1.00 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 5: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 5]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.90, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.13, 95% CI 2-sided [-2.23 to 1.97], Standard Error of Mean 1.07 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 6: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 6]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.04, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 2.05, 95% CI 2-sided [0.13 to 3.97], Standard Error of Mean 0.98 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 7: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 7]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.64, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.67, 95% CI 2-sided [-2.14 to 3.48], Standard Error of Mean 1.43 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 8: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 8]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.92, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.15, 95% CI 2-sided [-2.91 to 3.20], Standard Error of Mean 1.56 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 9: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 9]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.11, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -2.25, 95% CI 2-sided [-5.02 to 0.52], Standard Error of Mean 1.41 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter

3. Primary Outcome: Worry About Harms From Smoking
Description: A single question measured on a continuous scale to assess strength of worry about harms from smoking (1="Not at all", worse outcome; 7="Extremely", better outcome), with average scores (range=1-7) estimated.
Time Frame: as for outcome 1
Population: Analyses include repeated observations collected from daily cigarette surveys. The number of participants in the analytic sample is slightly smaller for H5 (control=101; insert only=84; pictorial warnings only=88; insert + pictorial warnings=88) due to missing data from the baseline survey that provides information for the moderating variables.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Cigarette Packs (Control) | Cigarette Packs With Inserts Only | Cigarette Packs With Pictorial Warnings Only | Cigarette Packs With Inserts and Pictorial Warnings
Number analyzed (Participants) | 101 | 86 | 90 | 89
score on a scale | 4.34 (1.94) | 4.84 (1.74) | 4.46 (1.91) | 4.47 (1.75)
Statistical Analysis 1: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; These results are for the pre-specified H2 assessment (see Statistical Analysis Plan, Model 1), comparing groups that received pictorial warnings (pictorial warning only AND insert + pictorial warnings) with the groups that did not (insert only AND control). We expected that the outcome would be higher in the pictorial warning groups than in the no pictorial warning groups; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.57, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.33, 95% CI 2-sided [-1.48 to 0.82], Standard Error of Mean 0.59 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 2: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; These results are for the intended (but not correctly pre-specified) H5a assessment, which evaluates moderation of the pre-specified H2 assessment. We expected that the effect of pictorial warnings (averaged over insert) vs no pictorial warnings (averaged over insert) on the outcome would be stronger for higher vs lower self-efficacy (see Statistical Analysis Plan, Model 4); Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.39, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.97, 95% CI 2-sided [-3.22 to 1.27], Standard Error of Mean 1.14 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 3: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; These results are for the intended (but not correctly pre-specified) H5b assessment, which evaluates whether moderation of pictorial warnings effects would vary by whether the pictorial warnings included inserts or not. We expected that moderation effects of baseline self-efficacy would be larger for pictorial warnings only (vs control) than for pictorial warnings AND inserts (vs control) (see Statistical Analysis Plan, Model 4); Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.92, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.16, 95% CI 2-sided [-3.35 to 3.04], Standard Error of Mean 1.63 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter

4. Primary Outcome: Strength of Feeling About Smoking
Description: A single question measured on a continuous scale to assess strength of positive to negative feelings about smoking (1="very bad", better outcome; 7="very good", worse outcome), with average scores (range=1-7) estimated
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Cigarette Packs (Control) | Cigarette Packs With Inserts Only | Cigarette Packs With Pictorial Warnings Only | Cigarette Packs With Inserts and Pictorial Warnings
Number analyzed (Participants) | 101 | 86 | 90 | 89
score on a scale | 3.98 (1.77) | 3.75 (1.60) | 3.71 (1.65) | 3.85 (1.67)
Statistical Analysis 1: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 3, analysis 1]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.40, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.40, 95% CI 2-sided [-1.33 to 0.53], Standard Error of Mean 0.48 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 2: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; These results are for the intended (but not correctly pre-specified) H5a assessment, which evaluates moderation of the pre-specified H2 assessment. We expected that the effect of pictorial health warning labels (HWLs) (averaged over insert) vs no pictorial HWLs (averaged over insert) on the outcome would be stronger for higher vs lower self-efficacy (see Statistical Analysis Plan, Model 4); Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.99, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.01, 95% CI 2-sided [-1.83 to 1.86], Standard Error of Mean 0.94 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 3: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 3, analysis 3]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.17, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 1.85, 95% CI 2-sided [-0.78 to 4.48], Standard Error of Mean 1.34 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter

5. Primary Outcome: Extent of Motivation to Quit Smoking
Description: A single question measured on a continuous scale to assess the extent of motivation to quit smoking (1="Not at all", worse outcome; 7="Extremely", better outcome), with average scores (range=1-7) estimated.
Time Frame: as for outcome 1
Population: Analyses include repeated observations from daily cigarette surveys. Due to missing data on moderators, the analytic sample differs for H5 (control=101; insert only=84; pictorial warnings only=88; insert + pictorial warnings=88) and for each H6 moderating variable: education (n=101, 84, 87, and 88, respectively); health literacy (n=101, 86, 90, and 88, respectively); and delayed discounting (n=101, 84, 88, and 88, respectively).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Cigarette Packs (Control) | Cigarette Packs With Inserts Only | Cigarette Packs With Pictorial Warnings Only | Cigarette Packs With Inserts and Pictorial Warnings
Number analyzed (Participants) | 101 | 86 | 90 | 89
score on a scale | 3.63 (1.64) | 4.00 (1.76) | 3.76 (1.79) | 3.62 (1.74)
Statistical Analysis 1: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 1]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.45, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.44, 95% CI 2-sided [-0.69 to 1.57], Standard Error of Mean 0.58 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 2: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 3, analysis 1]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.41, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.48, 95% CI 2-sided [-1.61 to 0.66], Standard Error of Mean 0.58 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 3: Comparison: Cigarette Packs With Inserts Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 2]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.08, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -1.44, 95% CI 2-sided [-3.08 to 0.20], Standard Error of Mean 0.84 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 4: Comparison: Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 3]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.52, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.52, 95% CI 2-sided [-2.14 to 1.09], Standard Error of Mean 0.82 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 5: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; These results are for the intended (but not correctly pre-specified) H5a assessment, which evaluates moderation of the pre-specified H2 assessment. We expected that the effect of pictorial HWLs (averaged over insert) vs no pictorial HWLs (averaged over insert) on the outcome would be stronger for higher vs lower self-efficacy (see Statistical Analysis Plan, Model 4); Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.75, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.35, 95% CI 2-sided [-1.82 to 2.51], Standard Error of Mean 1.11 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 6: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 3, analysis 3]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.64, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.74, 95% CI 2-sided [-3.82 to 2.33], Standard Error of Mean 1.57 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 7: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 4]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.91, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.14, 95% CI 2-sided [-2.17 to 2.45], Standard Error of Mean 1.18 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 8: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 5]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.50, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.84, 95% CI 2-sided [-3.29 to 1.60], Standard Error of Mean 1.25 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 9: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 6]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.007, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 3.14, 95% CI 2-sided [0.86 to 5.41], Standard Error of Mean 1.16 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 10: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 7]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.52, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 1.09, 95% CI 2-sided [-2.22 to 4.40], Standard Error of Mean 1.69 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 11: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 8]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.86, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.33, 95% CI 2-sided [-3.89 to 3.23], Standard Error of Mean 1.82 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 12: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 9]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.61, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.86, 95% CI 2-sided [-4.15 to 2.43], Standard Error of Mean 1.68 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter

6. Primary Outcome: Talk About Smoking Cessation
Description: For each day, a single binary variable was derived to indicate whether the participant talked about either smoking cessation or smoking-related harms in the prior 24 hours, with the average daily percentage of this outcome estimated. Experiencing the event of talking about cessation or harms is a better outcome, as it is a predictor of cessation attempts.
Time Frame: Evaluated once each day (evening survey) over the 14 day study period, with analyses limited to days 2-14. Day 1 was dropped due to varying intervention exposure and coverage of the day, depending on study orientation time.
Population: Analyses include repeated observations from evening reports. Due to missing data on moderators, the analytic sample differs for H5 (control=101; insert only=84; pictorial warnings only=88; insert + pictorial warnings=88) and for each H6 moderating variable: education (n=101, 85, 87, and 88, respectively); health literacy (n=101, 87, 90, and 88, respectively); and delayed discounting (n=101, 85, 88, and 88, respectively).
Measure: Mean (Standard Deviation); unit: percentage of days (events/days)
Arm/Group | Standard Cigarette Packs (Control) | Cigarette Packs With Inserts Only | Cigarette Packs With Pictorial Warnings Only | Cigarette Packs With Inserts and Pictorial Warnings
Number analyzed (Participants) | 101 | 87 | 90 | 88
percentage of days (events/days) | 0.1589 (0.3658) | 0.1645 (0.3709) | 0.1833 (0.3871) | 0.1898 (0.3924)
Statistical Analysis 1: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 1]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.29, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 1.26, 95% CI 2-sided [0.82 to 1.96], Standard Error of Mean 0.28 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 2: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 3, analysis 1]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.43, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.77 to 1.85], Standard Error of Mean 0.27 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 3: Comparison: Cigarette Packs With Inserts Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 2]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.60, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.63 to 2.20], Standard Error of Mean 0.37 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 4: Comparison: Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 3]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.48, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.67 to 2.33], Standard Error of Mean 0.40 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 5: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 5, analysis 5]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.62, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 0.80, 95% CI 2-sided [0.34 to 1.91], Standard Error of Mean 0.36 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 6: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 3, analysis 3]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.079, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 3.04, 95% CI 2-sided [0.88 to 10.52], Standard Error of Mean 1.93 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 7: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 4]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.10, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 2.10, 95% CI 2-sided [0.87 to 5.12], Standard Error of Mean 0.95 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 8: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 5]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.52, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 1.38, 95% CI 2-sided [0.52 to 3.61], Standard Error of Mean 0.68 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 9: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 6]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.54, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.55 to 3.17], Standard Error of Mean 0.59 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 10: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 7]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.33, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 1.88, 95% CI 2-sided [0.53 to 6.61], Standard Error of Mean 1.21 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 11: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 8]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.55, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 1.53, 95% CI 2-sided [0.38 to 6.11], Standard Error of Mean 1.08 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 12: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 9]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.44, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 0.61, 95% CI 2-sided [0.18 to 2.14], Standard Error of Mean 0.39 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 13: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; These results are for the multiple imputation models for pre-specified H1 assessment (see Statistical Analysis Plan, Model 1), comparing groups that received inserts (insert only AND insert + pictorial warnings) with the groups that did not (pictorial warning only AND control). We expected that the outcome would be higher in the insert groups than in the no insert groups; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.2510, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 1.29, 95% CI 2-sided [0.84 to 1.98], Standard Error of Mean 0.28 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 14: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; These results are for the multiple imputation model for the pre-specified H2 assessment (see Statistical Analysis Plan, Model 1), comparing groups that received pictorial warnings (pictorial warning only AND insert + pictorial warnings) with the groups that did not (insert only AND control). We expected that the outcome would be higher in the pictorial warning groups than in the no pictorial warning groups; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.2822, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.82 to 1.95], Standard Error of Mean 0.28 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 15: Comparison: Cigarette Packs With Inserts Only vs Cigarette Packs With Inserts and Pictorial Warnings; These results are for multiple imputation models for the pre-specified H3 assessment (see Statistical Analysis Plan, Model 1), comparing the group that received inserts and pictorial warnings with the group that received inserts only. We expected that this outcome would be higher in the insert and pictorial warning group than in the insert only group; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.3558, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 1.34, 95% CI 2-sided [0.72 to 2.47], Standard Error of Mean 0.42 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 16: Comparison: Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; These results are for the multiple imputation model for the pre-specified H4 assessment (see Statistical Analysis Plan, Model 1), comparing the group that received inserts and pictorial warnings with the group that received pictorial warnings only. We expected that this outcome would be higher in the insert and pictorial warning group than in the pictorial warning only group; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.3291, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 1.36, 95% CI 2-sided [0.73 to 2.51], Standard Error of Mean 0.43 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 17: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; These results are from the multiple imputation model for the intended (but not correctly pre-specified) H5a assessment, which evaluates moderation of the pre-specified H2 assessment. We expected that the effect of pictorial HWLs (averaged over insert) vs no pictorial HWLs (averaged over insert) on the outcome would be stronger for higher vs lower self-efficacy (see Statistical Analysis Plan, Model 4); Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.7818, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.38 to 2.09], Standard Error of Mean 0.39 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 18: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; These results are from the multiple imputation model for the intended (but not correctly pre-specified) H5b assessment, which evaluates whether moderation of pictorial warnings effects would vary by whether the pictorial warnings included inserts or not. We expected that moderation effects of baseline self-efficacy would be larger for pictorial warnings only (vs control) than for pictorial warnings AND inserts (vs control) (see Statistical Analysis Plan, Model 4); Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.0912, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 2.87, 95% CI 2-sided [0.84 to 9.73], Standard Error of Mean 1.79 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 19: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; These results are from the multiple imputation model for the intended (but not correctly pre-specified) H6a assessment, which evaluates moderation of the pre-specified H1 assessment. We expected that the effect of inserts (averaged over pictorial warnings) compared to no inserts (averaged over pictorial warnings) on the outcome would be stronger for those with higher than lower education (see Statistical Analysis Plan, Model 5); Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.1361, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 1.94, 95% CI 2-sided [0.81 to 4.66], Standard Error of Mean 0.87 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 20: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; These results are for the multiple imputation model for the intended (but not correctly pre-specified) H6a assessment, which evaluates moderation of the pre-specified H1 assessment. We expected that the effect of inserts (averaged over pictorial warnings) compared to no inserts (averaged over pictorial warnings) on the outcome would be stronger for those with higher than lower literacy (see Statistical Analysis Plan, Model 5); Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.7200, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.46 to 3.07], Standard Error of Mean 0.58 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 21: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; These results are from the multiple imputation model for the intended (but not correctly pre-specified) H6a assessment, which evaluates moderation of the pre-specified H1 assessment. We expected that the effect of inserts (averaged over pictorial warnings) compared to no inserts (averaged over pictorial warnings) on the outcome would be stronger for those with lower than higher delayed discounting (see Statistical Analysis Plan, Model 5); Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.3737, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 1.48, 95% CI 2-sided [0.62 to 3.53], Standard Error of Mean 0.66 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 22: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Inserts and Pictorial Warnings; These results are from the multiple imputation model for the intended (but not correctly pre-specified) H6b assessment, which evaluated whether the moderation of insert effects would vary by whether the inserts included pictorial warnings or not. We expected that moderation by baseline education would be stronger for insert only (vs control) than for inserts AND pictorial warnings (vs control) (see Statistical Analysis Plan, Model 5); Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.1345, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 2.58, 95% CI 2-sided [0.75 to 8.90], Standard Error of Mean 1.63 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 23: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Inserts and Pictorial Warnings; These results are from the multiple imputation model for the intended (but not correctly pre-specified) H6b assessment, which evaluated whether the moderation of insert effects would vary by whether the inserts included pictorial warnings or not. We expected that moderation by baseline literacy would be larger for insert only (vs control) than for inserts AND pictorial warnings (vs control) (see Statistical Analysis Plan, Model 5); Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.3318, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 1.96, 95% CI 2-sided [0.50 to 7.67], Standard Error of Mean 1.36 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 24: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Inserts and Pictorial Warnings; These results are from the multiple imputation model for the intended (but not correctly pre-specified) H6b assessment, which evaluated whether the moderation of insert effects would vary by whether the inserts included pictorial warnings or not. We expected that moderation by baseline delay discounting would be larger for insert only (vs control) than for inserts AND pictorial warnings (vs control) (see Statistical Analysis Plan, Model 5); Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.7017, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.23 to 2.70], Standard Error of Mean 0.49 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter

7. Primary Outcome: Foregoing a Cigarette
Description: For each day, responses to two questions were combined to create a binary variable for whether, in the prior 24 hours, the participant a) did not smoke a cigarette when they normally would, and/or b) stubbed out a cigarette before finishing it, with the average daily percentage of this outcome estimated. Experiencing the event of forgoing/stubbing out is a better outcome, as it is a predictor of cessation attempts.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Mean (Standard Error); unit: percentage of days (events/days)
Arm/Group | Standard Cigarette Packs (Control) | Cigarette Packs With Inserts Only | Cigarette Packs With Pictorial Warnings Only | Cigarette Packs With Inserts and Pictorial Warnings
Number analyzed (Participants) | 101 | 87 | 90 | 88
percentage of days (events/days) | 0.3882 (0.4876) | 0.5479 (0.498) | 0.4916 (0.5002) | 0.5807 (0.4937)
Statistical Analysis 1: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 1]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 2.47, 95% CI 2-sided [1.42 to 4.31], Standard Error of Mean 0.70 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 2: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 3, analysis 1]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.025, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 1.89, 95% CI 2-sided [1.09 to 3.30], Standard Error of Mean 0.54 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 3: Comparison: Cigarette Packs With Inserts Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 2]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.44, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 1.37, 95% CI 2-sided [0.62 to 3.06], Standard Error of Mean 0.56 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 4: Comparison: Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 3]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.15, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 1.80, 95% CI 2-sided [0.81 to 3.97], Standard Error of Mean 0.73 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 5: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 5, analysis 5]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.76, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.39 to 3.58], Standard Error of Mean 0.67 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 6: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 3, analysis 3]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.77, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.16 to 3.80], Standard Error of Mean 0.63 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 7: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 4]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.17, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 2.18, 95% CI 2-sided [0.72 to 6.61], Standard Error of Mean 1.23 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 8: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 5]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.22, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 0.46, 95% CI 2-sided [0.14 to 1.57], Standard Error of Mean 0.29 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 9: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 6]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.02, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 3.45, 95% CI 2-sided [1.15 to 10.37], Standard Error of Mean 1.94 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 10: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 7]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.04, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 5.45, 95% CI 2-sided [1.12 to 26.53], Standard Error of Mean 4.40 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 11: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 8]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.56, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 0.59, 95% CI 2-sided [0.10 to 3.47], Standard Error of Mean 0.53 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 12: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 9]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.46, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 0.55, 95% CI 2-sided [0.11 to 2.68], Standard Error of Mean 0.44 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 13: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; These results are from the multiple imputation model for the pre-specified H1 assessment (see Statistical Analysis Plan, Model 1), comparing groups that received inserts (insert only AND insert + pictorial warnings) with the groups that did not (pictorial warning only AND control). We expected that the outcome would be higher in the insert groups than in the no insert groups; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.0002, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 2.58, 95% CI 2-sided [1.56 to 4.27], Standard Error of Mean 0.66 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 14: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; These results are from the multiple imputation model for the pre-specified H2 assessment (see Statistical Analysis Plan, Model 1), comparing groups that received pictorial warnings (pictorial warning only AND insert + pictorial warnings) with the groups that did not (insert only AND control). We expected that the outcome would be higher in the pictorial warning groups than in the no pictorial warning groups; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.0135, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 1.89, 95% CI 2-sided [1.14 to 3.12], Standard Error of Mean 0.48 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 15: Comparison: Cigarette Packs With Inserts Only vs Cigarette Packs With Inserts and Pictorial Warnings; These results are from the multiple imputation model for the pre-specified H3 assessment (see Statistical Analysis Plan, Model 1), comparing the group that received inserts and pictorial warnings with the group that received inserts only. We expected that this outcome would be higher in the insert and pictorial warning group than in the insert only group; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.2619, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 1.51, 95% CI 2-sided [0.73 to 3.12], Standard Error of Mean 0.56 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 16: Comparison: Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; These results are from the multiple imputation model for the pre-specified H4 assessment (see Statistical Analysis Plan, Model 1), comparing the group that received inserts and pictorial warnings with the group that received pictorial warnings only. We expected that this outcome would be higher in the insert and pictorial warning group than in the pictorial warning only group; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.0474, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 2.07, 95% CI 2-sided [1.01 to 4.24], Standard Error of Mean 0.76 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 17: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 6, analysis 17]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.8094, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.42 to 3.07], Standard Error of Mean 0.58 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 18: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 6, analysis 18]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.7978, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 0.83, 95% CI 2-sided [0.20 to 3.44], Standard Error of Mean 0.60 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 19: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 6, analysis 19]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.1016, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 2.29, 95% CI 2-sided [0.85 to 6.15], Standard Error of Mean 1.15 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 20: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; These results are from the multiple imputation model for the intended (but not correctly pre-specified) H6a assessment, which evaluates moderation of the pre-specified H1 assessment. We expected that the effect of inserts (averaged over pictorial warnings) compared to no inserts (averaged over pictorial warnings) on the outcome would be stronger for those with higher than lower literacy (see Statistical Analysis Plan, Model 5); Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.1570, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 0.45, 95% CI 2-sided [0.15 to 1.36], Standard Error of Mean 0.25 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 21: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 6, analysis 21]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.0297, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 3.02, 95% CI 2-sided [1.11 to 8.18], Standard Error of Mean 1.53 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 22: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 6, analysis 22]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.0213, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 5.28, 95% CI 2-sided [1.28 to 21.73], Standard Error of Mean 3.81 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 23: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 6, analysis 23]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.9648, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.20 to 4.74], Standard Error of Mean 0.78 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 24: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Inserts and Pictorial Warnings; These results from the multiple imputation model are for the intended (but not correctly pre-specified) H6b assessment, which evaluated whether the moderation of insert effects would vary by whether the inserts included pictorial warnings or not. We expected that moderation by baseline delay discounting would be larger for insert only (vs control) than for inserts AND pictorial warnings (vs control) (see Statistical Analysis Plan, Model 5); Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.6512, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 0.72, Standard Error of Mean 0.53 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter

8. Secondary Outcome: Strength of Hopefulness About Quitting
Description: A single question measured on a continuous scale to assess strength of feeling hopeful about quitting (1="Not at all", worse outcome; 7="Extremely", better outcome), with average scores (range 1-7) estimated.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Cigarette Packs (Control) | Cigarette Packs With Inserts Only | Cigarette Packs With Pictorial Warnings Only | Cigarette Packs With Inserts and Pictorial Warnings
Number analyzed (Participants) | 101 | 86 | 90 | 89
score on a scale | 3.80 (1.80) | 4.25 (1.91) | 3.96 (1.87) | 3.86 (1.889)
Statistical Analysis 1: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 1]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.41, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.55, 95% CI 2-sided [-0.75 to 1.85], Standard Error of Mean 0.66 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 2: Comparison: Cigarette Packs With Inserts Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 2]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.08, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -1.67, 95% CI 2-sided [-3.55 to 0.21], Standard Error of Mean 0.96 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 3: Comparison: Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 3]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.55, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.57, 95% CI 2-sided [-2.42 to 1.29], Standard Error of Mean 0.95 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 4: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 4]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.38, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 1.20, 95% CI 2-sided [-1.47 to 3.86], Standard Error of Mean 1.36 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 5: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 5]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.71, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.54, 95% CI 2-sided [-3.35 to 2.28], Standard Error of Mean 1.44 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 6: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 6]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.02, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 3.21, 95% CI 2-sided [0.59 to 5.83], Standard Error of Mean 1.34 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 7: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 7]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.98, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.05, 95% CI 2-sided [-3.85 to 3.76], Standard Error of Mean 1.94 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 8: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 8]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.31, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -2.13, 95% CI 2-sided [-6.2 to 1.95], Standard Error of Mean 2.08 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 9: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 9]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.68, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.8, 95% CI 2-sided [-4.58 to 2.97], Standard Error of Mean 1.93 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter

9. Secondary Outcome: Extent of Cognitive Elaboration of Smoking Benefits
Description: A single question measured on a continuous scale to assess the frequency of thinking about the positive things about smoking (1="Not at all", better outcome; 7="Extremely", worse outcome), with average scores (range 1-7) estimated.
Time Frame: as for outcome 6
Population: Analyses include repeated observations collected from evening surveys.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Cigarette Packs (Control) | Cigarette Packs With Inserts Only | Cigarette Packs With Pictorial Warnings Only | Cigarette Packs With Inserts and Pictorial Warnings
Number analyzed (Participants) | 101 | 86 | 89 | 89
score on a scale | 3.19 (1.72) | 3.20 (1.64) | 3.16 (1.69) | 3.17 (1.70)
Statistical Analysis 1: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 3, analysis 1]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.45, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects ordered logistic regression models that accounted for repeated measures at the individual level; Mean Difference (Net) = -0.23, 95% CI 2-sided [-0.81 to 0.36], Standard Error of Mean 0.30 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 2: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; These results from the multiple imputation model are for the pre-specified H2 assessment (see Statistical Analysis Plan, Model 1), comparing groups that received pictorial warnings (pictorial warning only AND insert + pictorial warnings) with the groups that did not (insert only AND control). We expected that the outcome would be higher in the pictorial warning groups than in the no pictorial warning groups; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.5767, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = -0.14, 95% CI 2-sided [-0.64 to 0.70], Standard Error of Mean 0.25 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter

10. Secondary Outcome: Extent of Cognitive Elaboration of Smoking Harms
Description: A single question measured on a continuous scale to assess the frequency of thinking about the harms from smoking (1="Not at all", worse outcome; 7="Extremely", better outcome), with average scores (range 1-7) estimated.
Time Frame: as for outcome 6
Population: Analyses include repeated observations collected from daily cigarette surveys or evening reports, depending on the outcome. The number of participants in the analytic sample is slightly smaller for H5 (control=101; insert only=84; pictorial warnings only=88; insert + pictorial warnings=88) due to missing data from the baseline survey that provides information for the moderating variables.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Cigarette Packs (Control) | Cigarette Packs With Inserts Only | Cigarette Packs With Pictorial Warnings Only | Cigarette Packs With Inserts and Pictorial Warnings
Number analyzed (Participants) | 101 | 87 | 89 | 89
score on a scale | 3.91 (1.83) | 4.40 (1.77) | 3.95 (1.89) | 4.15 (1.77)
Statistical Analysis 1: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 3, analysis 1]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.36, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = -0.31, 95% CI 2-sided [-0.98 to 0.36], Standard Error of Mean 0.34 — We estimated mixed-effects ordered logistic regression models that accounted for repeated measures at the individual level
Statistical Analysis 2: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 5, analysis 5]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.63, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = -0.32, 95% CI 2-sided [-1.64 to 0.99], Standard Error of Mean 0.67 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 3: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 3, analysis 3]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.79, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = 0.25, 95% CI 2-sided [-1.62 to 2.12], Standard Error of Mean 0.95 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 4: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 9, analysis 2]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.4491, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = -0.23, 95% CI 2-sided [-0.84 to 0.37], Standard Error of Mean 0.31 — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 5: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; These results from the multiple imputation model are for the intended (but not correctly pre-specified) H5a assessment, which evaluates moderation of the pre-specified H2 assessment. We expected that the effect of pictorial HWLs (averaged over insert) vs no pictorial HWLs (averaged over insert) on the outcome would be stronger for higher vs lower self-efficacy (see Statistical Analysis Plan, Model 4); Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.8713, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = -0.10, 95% CI 2-sided [-1.26 to 1.06], Standard Error of Mean 0.59 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 6: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; These results from the multiple imputation model are for the intended (but not correctly pre-specified) H5b assessment, which evaluates whether moderation of pictorial warnings effects would vary by whether the pictorial warnings included inserts or not. We expected that moderation effects of baseline self-efficacy would be larger for pictorial warnings only (vs control) than for pictorial warnings AND inserts (vs control) (see Statistical Analysis Plan, Model 4); Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.99, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = 0.00, 95% CI 2-sided [-1.66 to 1.66], Standard Error of Mean 0.85 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter

11. Secondary Outcome: Extent of Cognitive Elaboration of Cessation Benefits
Description: A single question measured on a continuous scale to assess the frequency of thinking about the potential benefits from cessation (1="Not at all", worse outcome; 7="Extremely", better outcome), with average scores (range 1-7) estimated.
Time Frame: as for outcome 6
Population: Analyses include repeated observations from evening reports. Analytic samples for H6 differ due to some missing data for each moderating variable: education (control=101; insert only=84; pictorial warnings only=87; insert + pictorial warnings=88); health literacy (control=101; insert only=86; pictorial warnings only=90; insert + pictorial warnings=88); and delayed discounting (control=101; insert only=84; pictorial warnings only=88; insert + pictorial warnings=88).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Cigarette Packs (Control) | Cigarette Packs With Inserts Only | Cigarette Packs With Pictorial Warnings Only | Cigarette Packs With Inserts and Pictorial Warnings
Number analyzed (Participants) | 101 | 86 | 89 | 89
score on a scale | 4.07 (1.81) | 4.62 (1.77) | 4.13 (1.90) | 4.34 (1.77)
Statistical Analysis 1: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 1]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.04, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = 0.69, 95% CI 2-sided [0.02 to 1.37], Standard Error of Mean 0.34 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 2: Comparison: Cigarette Packs With Inserts Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 2]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.08, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = -0.87, 95% CI 2-sided [-1.85 to 0.11], Standard Error of Mean 0.50 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 3: Comparison: Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 3]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.65, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = 0.23, 95% CI 2-sided [-0.74 to 1.19], Standard Error of Mean 0.49 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 4: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 4]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.30, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = 0.73, 95% CI 2-sided [-0.66 to 2.11], Standard Error of Mean 0.71 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 5: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 5]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.78, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = -0.21, 95% CI 2-sided [-1.68 to 1.26], Standard Error of Mean 0.75 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 6: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 6]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.03, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = 1.48, 95% CI 2-sided [0.12 to 2.83], Standard Error of Mean 0.69 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 7: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 7]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.95, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = 0.06, 95% CI 2-sided [-1.92 to 2.04], Standard Error of Mean 1.01 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 8: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 8]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.48, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = -0.78, 95% CI 2-sided [-2.91 to 1.36], Standard Error of Mean 1.09 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 9: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 9]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.37, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = -0.90, 95% CI 2-sided [-2.86 to 1.07], Standard Error of Mean 1.00 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 10: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; These results from the multiple imputation model are for the pre-specified H1 assessment (see Statistical Analysis Plan, Model 1), comparing groups that received inserts (insert only AND insert + pictorial warnings) with the groups that did not (pictorial warning only AND control). We expected that the outcome would be higher in the insert groups than in the no insert groups; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.0192, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = 0.73, 95% CI 2-sided [0.12 to 1.34], Standard Error of Mean 0.31 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 11: Comparison: Cigarette Packs With Inserts Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 7, analysis 15]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.1860, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = -0.59, 95% CI 2-sided [-1.48 to 0.29], Standard Error of Mean 0.45 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 12: Comparison: Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; These results from the multiple imputation model are for the pre-specified H4 assessment (see Statistical Analysis Plan, Model 1), comparing the group that received inserts and pictorial warnings with the group that received pictorial warnings only. We expected that this outcome would be higher in the insert and pictorial warning group than in the pictorial warning only group; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.3863, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = 0.39, 95% CI 2-sided [-0.49 to 1.26], Standard Error of Mean 0.44 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 13: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; These results from the multiple imputation model are for the intended (but not correctly pre-specified) H6a assessment, which evaluates moderation of the pre-specified H1 assessment. We expected that the effect of inserts (averaged over pictorial warnings) compared to no inserts (averaged over pictorial warnings) on the outcome would be stronger for those with higher than lower education (see Statistical Analysis Plan, Model 5); Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.5710, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = 0.36, 95% CI 2-sided [-0.89 to 1.61], Standard Error of Mean 0.64 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 14: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; These results from the multiple imputation model are for the intended (but not correctly pre-specified) H6a assessment, which evaluates moderation of the pre-specified H1 assessment. We expected that the effect of inserts (averaged over pictorial warnings) compared to no inserts (averaged over pictorial warnings) on the outcome would be stronger for those with higher than lower literacy (see Statistical Analysis Plan, Model 5); Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.2797, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = -0.73, 95% CI 2-sided [-2.06 to 0.60], Standard Error of Mean 0.68 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 15: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; These results from the multiple imputation model are for the intended (but not correctly pre-specified) H6a assessment, which evaluates moderation of the pre-specified H1 assessment. We expected that the effect of inserts (averaged over pictorial warnings) compared to no inserts (averaged over pictorial warnings) on the outcome would be stronger for those with lower than higher delayed discounting (see Statistical Analysis Plan, Model 5); Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.0312, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = 1.33, 95% CI 2-sided [0.12 to 2.55], Standard Error of Mean 0.62 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 16: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Inserts and Pictorial Warnings; These results from the multiple imputation model are for the intended (but not correctly pre-specified) H6b assessment, which evaluated whether the moderation of insert effects would vary by whether the inserts included pictorial warnings or not. We expected that moderation by baseline education would be stronger for insert only (vs control) than for inserts AND pictorial warnings (vs control) (see Statistical Analysis Plan, Model 5); Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.5086, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = 0.60, 95% CI 2-sided [-1.19 to 2.39], Standard Error of Mean 0.91 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 17: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 6, analysis 23]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.9474, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = 0.06, 95% CI 2-sided [-1.86 to 1.99], Standard Error of Mean 0.98 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 18: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 7, analysis 24]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.5018, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = -0.60, 95% CI 2-sided [-2.36 to 1.16], Standard Error of Mean 0.90 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter

12. Secondary Outcome: Strength of Beliefs About Benefits of Smoking Cessation (i.e., Response Efficacy)
Description: A single question measured on a continuous scale to assess the strength of perceived benefits from cessation (1="Not at all", worse outcome; 7="Extremely", better outcome), with average scores (range 1-7) estimated.
Time Frame: as for outcome 6
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Standard Cigarette Packs (Control) | Cigarette Packs With Inserts Only | Cigarette Packs With Pictorial Warnings Only | Cigarette Packs With Inserts and Pictorial Warnings
Number analyzed (Participants) | 101 | 87 | 89 | 89
Score on a scale | 4.69 (1.87) | 5.18 (1.51) | 4.96 (1.78) | 4.95 (1.65)
Statistical Analysis 1: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 1]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.25, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = 0.45, 95% CI 2-sided [-0.31 to 1.21], Standard Error of Mean 0.39 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 2: Comparison: Cigarette Packs With Inserts Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 2]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.34, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = -0.53, 95% CI 2-sided [-1.63 to 0.57], Standard Error of Mean 0.56 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 3: Comparison: Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 3]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.76, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = -0.17, 95% CI 2-sided [-1.26 to 0.92], Standard Error of Mean 0.56 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 4: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 4]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.15, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = 1.10, 95% CI 2-sided [-0.42 to 2.63], Standard Error of Mean 0.78 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 5: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 5]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 1.00, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = -0.003, 95% CI 2-sided [-1.66 to 1.66], Standard Error of Mean 0.85 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 6: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 6]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.01, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = 1.90, 95% CI 2-sided [0.38 to 3.43], Standard Error of Mean 0.78 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 7: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 7]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.58, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = 0.62, 95% CI 2-sided [-1.56 to 2.80], Standard Error of Mean 1.11 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 8: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 8]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.39, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = -1.06, 95% CI 2-sided [-3.47 to 1.35], Standard Error of Mean 1.23 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 9: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 9]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.45, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = -0.85, 95% CI 2-sided [-3.05 to 1.35], Standard Error of Mean 1.12 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 10: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 11, analysis 10]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.1147, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = 0.54, 95% CI 2-sided [-0.13 to 1.21], Standard Error of Mean 0.34 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 11: Comparison: Cigarette Packs With Inserts Only vs Cigarette Packs With Inserts and Pictorial Warnings; These results from the multiple imputation model are for the pre-specified H3 assessment (see Statistical Analysis Plan, Model 1), comparing the group that received inserts and pictorial warnings with the group that received inserts only. We expected that this outcome would be higher in the insert and pictorial warning group than in the insert only group; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.3721, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = -0.44, 95% CI 2-sided [-1.41 to 0.53], Standard Error of Mean 0.49 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 12: Comparison: Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 7, analysis 16]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.8827, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = 0.07, 95% CI 2-sided [-0.89 to 1.03], Standard Error of Mean 0.49 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 13: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 11, analysis 13]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.4335, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = 0.54, 95% CI 2-sided [-0.80 to 1.87], Standard Error of Mean 0.68 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 14: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 7, analysis 20]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.4063, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = -0.62, 95% CI 2-sided [-2.07 to 0.84], Standard Error of Mean 0.74 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 15: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 11, analysis 15]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.0132, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = 1.69, 95% CI 2-sided [0.35 to 3.03], Standard Error of Mean 0.68 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 16: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 11, analysis 16]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.3949, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = 0.83, 95% CI 2-sided [-1.08 to 2.75], Standard Error of Mean 0.98 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 17: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Inserts and Pictorial Warnings; These results from the multiple imputation model are for the intended (but not correctly pre-specified) H6b assessment, which evaluated whether the moderation of insert effects would vary by whether the inserts included pictorial warnings or not. We expected that moderation by baseline literacy would be larger for insert only (vs control) than for inserts AND pictorial warnings (vs control) (see Statistical Analysis Plan, Model 5); Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.7145, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = -0.39, 95% CI 2-sided [-2.50 to 1.72], Standard Error of Mean 1.08 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 18: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 7, analysis 24]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.6081, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = -0.51, Standard Error of Mean 0.98 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter

13. Secondary Outcome: Strength of Perceived Susceptibility to Smoking Harms
Description: A single question measured on a continuous scale to assess the perceived likelihood of suffering harms from smoking (1="Not at all", worse outcome; 7="Extremely", better outcome), with average scores (range 1-7) estimated.
Time Frame: as for outcome 6
Population: Analyses include repeated observations collected from evening reports. The number of participants in the analytic sample is slightly smaller for H5 (control=101; insert only=84; pictorial warnings only=88; insert + pictorial warnings=88) due to missing data from the baseline survey that provides information for the moderating variable.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Cigarette Packs (Control) | Cigarette Packs With Inserts Only | Cigarette Packs With Pictorial Warnings Only | Cigarette Packs With Inserts and Pictorial Warnings
Number analyzed (Participants) | 101 | 87 | 89 | 89
score on a scale | 4.95 (1.81) | 5.53 (1.42) | 5.21 (1.76) | 5.21 (1.61)
Statistical Analysis 1: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 3, analysis 1]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.58, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = -0.26, 95% CI 2-sided [-1.15 to 0.64], Standard Error of Mean 0.46 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 2: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 5, analysis 5]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.82, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = -0.20, 95% CI 2-sided [-1.98 to 1.57], Standard Error of Mean 0.90 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 3: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 3, analysis 3]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.20, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = 1.67, 95% CI 2-sided [-0.90 to 4.24], Standard Error of Mean 1.31 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 4: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; These results from the multiple imputation analysis are for the pre-specified H2 assessment (see Statistical Analysis Plan, Model 1), comparing groups that received pictorial warnings (pictorial warning only AND insert + pictorial warnings) with the groups that did not (insert only AND control). We expected that the outcome would be higher in the pictorial warning groups than in the no pictorial warning groups; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.8800, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = -0.05, 95% CI 2-sided [-0.77 to 0.66], Standard Error of Mean 0.36 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 5: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 10, analysis 5]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.8864, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 9, analysis 1]; Median Difference (Net) = 0.10, 95% CI 2-sided [-1.30 to 1.50], Standard Error of Mean 0.72 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 6: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 10, analysis 6]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.2748, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = 1.12, 95% CI 2-sided [-0.89 to 3.12], Standard Error of Mean 1.02 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter

14. Secondary Outcome: Expressed Reactance Against Health Messages
Description: a. Binary measure for whether the participant reported talking about how health information on packs is either useless or not believable in the prior 24 hours, with the average daily percentage of this outcome estimated. Experiencing the event is a worse outcome, as it suggests defensive responding to labels.
Time Frame: as for outcome 6
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percentage of days (events/days)
Arm/Group | Standard Cigarette Packs (Control) | Cigarette Packs With Inserts Only | Cigarette Packs With Pictorial Warnings Only | Cigarette Packs With Inserts and Pictorial Warnings
Number analyzed (Participants) | 101 | 87 | 90 | 89
percentage of days (events/days) | 0.0103 (0.1011) | 0.0194 (0.1380) | 0.0369 (0.1885) | 0.0157 (0.1242)
Statistical Analysis 1: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; These results are for the pre-specified H1 assessment (see Statistical Analysis Plan, Model 1), comparing groups that received inserts (insert only AND insert + pictorial warnings) with the groups that did not (pictorial warning only AND control). We expected that the outcome would be lower in the insert groups than in the no insert groups; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.83, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.45 to 2.70], Standard Error of Mean 0.50 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 2: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 3, analysis 1]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.03, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 2.86, 95% CI 2-sided [1.14 to 7.18], Standard Error of Mean 1.34 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 3: Comparison: Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; These results are for the pre-specified H4 assessment (see Statistical Analysis Plan, Model 1), comparing the group that received inserts and pictorial warnings with the group that received pictorial warnings only. We expected that this outcome would be lower in the insert and pictorial warning group than in the pictorial warning only group; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.18, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 0.53, 95% CI 2-sided [0.15 to 1.44], Standard Error of Mean 0.27 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 4: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; These results are for the intended (but not correctly pre-specified) H5a assessment, which evaluates moderation of the pre-specified H2 assessment. We expected that the effect of pictorial HWLs (averaged over insert) vs no pictorial HWLs (averaged over insert) on the outcome would be lower for higher vs lower self-efficacy (see Statistical Analysis Plan, Model 4); Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.99, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.08 to 12.57], Standard Error of Mean 1.30 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 5: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 3, analysis 3]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.86, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.29 to 2.82], Standard Error of Mean 0.52
Statistical Analysis 6: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; These results from the multiple imputation model are for the pre-specified H1 assessment (see Statistical Analysis Plan, Model 1), comparing groups that received inserts (insert only AND insert + pictorial warnings) with the groups that did not (pictorial warning only AND control). We expected that the outcome would be lower in the insert groups than in the no insert groups; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.8045, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 1.10, Standard Error of Mean 0.43 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 7: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 7, analysis 14]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.0205, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 2.53, Standard Error of Mean 1.01 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 8: Comparison: Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; These results from the multiple imputation model are for the pre-specified H4 assessment (see Statistical Analysis Plan, Model 1), comparing the group that received inserts and pictorial warnings with the group that received pictorial warnings only. We expected that this outcome would be lower in the insert and pictorial warning group than in the pictorial warning only group; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.1918, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 0.53, Standard Error of Mean 0.26 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 9: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; These results are from the multiple imputation model for the intended (but not correctly pre-specified) H5a assessment, which evaluates moderation of the pre-specified H2 assessment. We expected that the effect of pictorial HWLs (averaged over insert) vs no pictorial HWLs (averaged over insert) on the outcome would be lower for higher vs lower self-efficacy (see Statistical Analysis Plan, Model 4); Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.99, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 1.03, Standard Error of Mean 1.12 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 10: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 6, analysis 18]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.6873, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; We estimated mixed-effects logistic regression models that accounted for repeated measures at the individual level; Odds Ratio (OR) = 1.56, Standard Error of Mean 1.54 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter

15. Secondary Outcome: Satisfaction From Smoking
Description: Single question measured on a continuous scale that assesses strength of satisfaction from smoking (1="Not at all", better outcome; 7="Extremely", worse outcome), with average scores (range 1-7) estimated.
Time Frame: as for outcome 1
Population: Analyses include repeated observations collected from daily cigarette surveys.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Cigarette Packs (Control) | Cigarette Packs With Inserts Only | Cigarette Packs With Pictorial Warnings Only | Cigarette Packs With Inserts and Pictorial Warnings
Number analyzed (Participants) | 101 | 86 | 90 | 89
score on a scale | 4.95 (1.47) | 4.89 (1.43) | 4.74 (1.56) | 4.83 (1.45)
Statistical Analysis 1: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 3, analysis 1]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.37, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.35, 95% CI 2-sided [-1.12 to 0.41], Standard Error of Mean 0.39 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter

16. Secondary Outcome: Cigarettes Logged
Description: Continuous variable summing the total number of cigarettes logged over the study period. Lower values represent a better outcome (i.e., fewer cigarettes smoked).
Time Frame: Participants logged each cigarette smoked over the 14 day study period, with analyses limited to reports from days 2-14. Day 1 and 15 were dropped due to varying coverage of the day depending on study orientation time (Day 1) and ending (Day 15).
Population: Analyses assess the sum of all cigarettes participants logged from days 2-14 of the study. Due to missing data on moderators, the analytic sample differs for H5 (control=101; insert only=84; pictorial warnings only=88; insert + pictorial warnings=88) and for each H6 moderating variable: education (n=101, 85, 87, and 88, respectively); health literacy (n=101, 87, 90, and 88, respectively); and delayed discounting (n=101, 85, 88, and 88, respectively).
Measure: Mean (Standard Deviation); unit: cigarettes
Arm/Group | Standard Cigarette Packs (Control) | Cigarette Packs With Inserts Only | Cigarette Packs With Pictorial Warnings Only | Cigarette Packs With Inserts and Pictorial Warnings
Number analyzed (Participants) | 101 | 87 | 90 | 89
cigarettes | 181.1 (81.90) | 185.9 (95.85) | 190.3 (103.00) | 185.8 (97.42)
Statistical Analysis 1: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 1]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.92, Negative binomial regression — [p-value comment as in outcome 1, analysis 1]; We estimated negative binomial regression models, as there is a single measure for each person and so there are no repeated measures; Rate ratio = 0.99, 95% CI 2-sided [0.90 to 1.10], Standard Error of Mean 0.05 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 2: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 3, analysis 1]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.95, Negative binomial regression — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 16, analysis 1]; Rate ratio = 1, 95% CI 2-sided [0.90 to 1.11], Standard Error of Mean 0.05 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 3: Comparison: Cigarette Packs With Inserts Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 2]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.85, Negative binomial regression — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 16, analysis 1]; Rate ratio = 0.99, 95% CI 2-sided [0.85 to 1.14], Standard Error of Mean 0.08 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 4: Comparison: Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 3]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.75, Negative binomial regression — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 16, analysis 1]; Rate ratio = 0.98, 95% CI 2-sided [0.84 to 1.13], Standard Error of Mean 0.07 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 5: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 5, analysis 5]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.78, Negative binomial regression — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 16, analysis 1]; Rate ratio = 0.97, 95% CI 2-sided [0.78 to 1.20], Standard Error of Mean 0.11 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 6: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 3, analysis 3]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.11, Negative binomial regression — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 16, analysis 1]; Rate ratio = 1.31, 95% CI 2-sided [0.94 to 1.82], Standard Error of Mean 0.22 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 7: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 4]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.93, Negative binomial regression — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 16, analysis 1]; Rate ratio = 0.99, 95% CI 2-sided [0.80 to 1.22], Standard Error of Mean 0.11 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 8: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 5]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.86, Negative binomial regression — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 16, analysis 1]; Rate ratio = 0.98, 95% CI 2-sided [0.78 to 1.23], Standard Error of Mean 0.11 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 9: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Pictorial Warnings Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 6]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.94, Negative binomial regression — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 16, analysis 1]; Rate ratio = 0.99, 95% CI 2-sided [0.81 to 1.22], Standard Error of Mean 0.11 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 10: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 7]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.13, Negative binomial regression — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 16, analysis 1]; Rate ratio = 1.29, 95% CI 2-sided [0.93 to 1.78], Standard Error of Mean 0.21 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 11: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 8]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.96, Negative binomial regression — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 16, analysis 1]; Rate ratio = 0.99, 95% CI 2-sided [0.70 to 1.41], Standard Error of Mean 0.18 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter
Statistical Analysis 12: Comparison: Standard Cigarette Packs (Control) vs Cigarette Packs With Inserts Only vs Cigarette Packs With Inserts and Pictorial Warnings; [analysis description as in outcome 1, analysis 9]; Test type: Other — We conducted a two-sided test for mean (group 1) = mean (group 2) versus means not being equal; p = 0.95, Negative binomial regression — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 16, analysis 1]; Rate ratio = 0.99, 95% CI 2-sided [0.72 to 1.36], Standard Error of Mean 0.16 — To evaluate the study hypothesis, a Wald test was used for the associated regression parameter

17. Other Pre Specified Outcome: Conversation Partners
Description: Nominal variable indicating the types of people with whom people talked about smoking and cessation in the prior 24 hours
Time Frame: as for outcome 6
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Conversation Topics
Description: Nominal variable indicating the topics of conversation around smoking in the prior 24 hours
Time Frame: as for outcome 6
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were assessed during the 14 day study participation period.
Description: Adverse events were detected through the standardized study protocol of phoning participants when they stopped recording cigarettes and responding to evening surveys. Through this approach, we detected two adverse events that required hospitalization and may have been caused by long-term smoking.
Arm/Group | Standard Cigarette Packs (Control) | Cigarette Packs With Inserts Only | Cigarette Packs With Pictorial Warnings Only | Cigarette Packs With Inserts and Pictorial Warnings
All-Cause Mortality (participants affected / at risk) | 0/108 | 0/94 | 0/94 | 0/91
Serious Adverse Events (participants affected / at risk) | 0/108 | 1/94 | 1/94 | 0/91
Other Adverse Events (participants affected / at risk) | 0/108 | 0/94 | 0/94 | 0/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Cigarette Packs (Control) (N=108) | Cigarette Packs With Inserts Only (N=94) | Cigarette Packs With Pictorial Warnings Only (N=94) | Cigarette Packs With Inserts and Pictorial Warnings (N=91)
Heart Attack (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — One participant in the inserts only condition was found to have been hospitalized after experiencing a heart attack when the study team followed up with him to determine why he had stopped logging cigarettes and surveys.
Mini stroke (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — One participant in the pictorial warning only group was found to have experienced what he termed a "mini stroke" when the study team followed up with him to determine why he had stopped logging cigarettes and surveys.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-06-23): https://cdn.clinicaltrials.gov/large-docs/82/NCT04075682/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-13): https://cdn.clinicaltrials.gov/large-docs/82/NCT04075682/SAP_001.pdf
  • Informed Consent Form (2020-07-21): https://cdn.clinicaltrials.gov/large-docs/82/NCT04075682/ICF_002.pdf